CLINICAL TRIAL: NCT05774132
Title: Ultrasound Guided Subgluteal Sciatic Nerve Block Versus Caudal Analgesia in Pediatric Patients With Spastic Cerebral Palsy Undergoing Lower Limb Multi-level Soft Tissue Corrective Surgeries
Brief Title: Ultrasound Guided Subgluteal Sciatic Nerve Block Versus Caudal Analgesia for Cerebral Palsy Patients Undergoing Lower Limb Corrective Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, hany magdy fahim, Lecturer of anesthesia , Intensive care and pain management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FMASU R24/ 2023
Record Dates: First submitted 2023-03-04; First posted 2023-03-17 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound guided Subgluteal sciatic nerve block group (Active Comparator): using 0.25% bupivacaine ( 0.3ml/Kg )
  Interventions: Procedure: ultrasound guided Subgluteal sciatic nerve block
- ultrasound guided Caudal block group (Active Comparator): using 0.25% bupivacaine ( 1ml/Kg)
  Interventions: Procedure: ultrasound guided Caudal block

INTERVENTIONS:
Procedure: ultrasound guided Subgluteal sciatic nerve block — Patients will be positioned in lateral decubitus and the ultrasound scanning for the sciatic nerve in the subgluteal region will be started between the two bony landmarks (greater trochanter and ischial tuberosity ) using high frequency linear probe then approached via 5 cm block needle under ultrasound guidance after which bupivacaine 0.25% (0.3 ml/kg) will be administered in increments .
  Arms: ultrasound guided Subgluteal sciatic nerve block group
Procedure: ultrasound guided Caudal block — Patients will be positioned in lateral decubitus and their sacral hiatus will be palpated under the scanning of the ultrasound using high frequency linear probe then approached via 5 cm block needle that pierce the sacrococcygeal ligament then will be advanced to caudal canal under ultrasound guidance after which bupivacaine 0.25% (1 ml/kg) will be administered in increments.
  Arms: ultrasound guided Caudal block group

SUMMARY:
Both caudal and peripheral nerve blocks are widely used for postoperative analgesia in pediatric population .The safety of both techniques has been documented especially after the application of ultrasound guidance for their performance. Patients with cerebral palsy usually require lower limb orthopedic surgeries,that extend from minor soft tissue releases, like tenotomies, tendon lengthening or transfer, to major osteotomies for correction of their limb deformities.

Study objective: to compare the efficacy of ultrasound guided caudal block with subgluteal sciatic nerve block for postoperative pain control in pediatric patients with cerebral palsy who will undergo soft tissue surgeries for knee and ankle deformities correction.

Methods: This study patients will be randomly distributed to 2 Groups to receive either US guided caudal block or US subgluteal sciatic nerve block after induction of general anesthesia.

DETAILED DESCRIPTION:
After proper preoperative patients' anesthesia assessment; the study patients (15 per each group) will receive general anesthesia with either intravenous induction or inhalational induction if uncooperative under full monitoring of hemodynamics, temperature and oxygen saturation.

In caudal group : Patients will be positioned in lateral decubitus and their sacral hiatus will be palpated under the scanning of the ultrasound using high frequency linear probe then approached via 5 cm block needle that pierce the sacrococcygeal ligament then will be advanced to caudal canal under ultrasound guidance after which Marcaine 0.25% (1 ml/kg) will be administered in increments.

In subgluteal sciatic group : Patients will be positioned in lateral decubitus and the ultrasound scanning for the sciatic nerve in the subgluteal region will be started between the two bony landmarks (greater trochanter and ischial tuberosity ) using high frequency linear probe then approached via 5 cm block needle under ultrasound guidance after which Marcaine 0.25% (0.3 ml/kg) will be administered in increments .

Anesthesia will be maintained with sevoflurane inhalational anesthesia and incremental rocuronium and fentanyl for muscle relaxation and intraoperative analgesia respectively . Muscle relaxation will be reversed at the end of surgery by atropine-neostigmine combination and patients will be extubated fully awake. Postoperative analgesia in the form of intravenous paracetamol 15 mg/kg will be administered if revised FLACC(face,legs,activity,cry and consolability) scores are ≥ 4 and intravenous infusion of ketorolac 0.5 mg/ kg will be given if pain persisted for 15 minutes after paracetamol injection

ELIGIBILITY:
Inclusion Criteria:

* Patient with spastic cerebral palsy
* Age 2 -12 years
* Both gender
* ASA ( American society of anesthesiologists) physical status II

Exclusion Criteria:

* Parents' refusal to study participation.
* Patients with dyskinetic or ataxic cerebral palsy
* Patients need surgery for hip contracture/deformity
* Severe mental dysfunction
* Poor controlled epilepsy
* Advanced respiratory,renal or hepatic impairment
* Allergy to study medications
* Block contraindication as skin infection near to the block site, gross deformities and bleeding disorders.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
The time till the first postoperative analgesia demand | within 24 hours after surgery

SECONDARY OUTCOMES:
Postoperative revised FLACC scores | 2 hours postoperative
  Revised FLACC score ( face,leg,activity, cry and consolability) score Behaviour 0 1 2 Face No particular expression or smile Occasional grimace or frown, withdrawn, disinterested Frequent to constant quivering chin, clenched jow Legs Normal position or relaxed Uneasy, restless, tense Kicking or legs drawn up Activity Lying quietly, normal position, moves easily Squirming, shifting, back and forth, tense Arched, rigid or jerking Cry No cry (awake or asleep) Moans or whimpers; occasional complaint Crying steadily, screams, sobs, frequent complaints Consolability Content, relaxed Reassured by touching, hugging or being talked to, distractible Difficult to console or comfort 0 = Relaxed and comfortable 1-3 = Mild discomfort 4-6 = Moderate pain 7-10 = Severe discomfort/pain
Postoperative revised FLACC scores | 4 hours postoperative
  Revised FLACC score ( face,leg,activity, cry and consolability) score Behaviour 0 1 2 Face No particular expression or smile Occasional grimace or frown, withdrawn, disinterested Frequent to constant quivering chin, clenched jow Legs Normal position or relaxed Uneasy, restless, tense Kicking or legs drawn up Activity Lying quietly, normal position, moves easily Squirming, shifting, back and forth, tense Arched, rigid or jerking Cry No cry (awake or asleep) Moans or whimpers; occasional complaint Crying steadily, screams, sobs, frequent complaints Consolability Content, relaxed Reassured by touching, hugging or being talked to, distractible Difficult to console or comfort 0 = Relaxed and comfortable 1-3 = Mild discomfort 4-6 = Moderate pain 7-10 = Severe discomfort/pain
Postoperative revised FLACC scores | 6 hours postoperative
  Revised FLACC score ( face,leg,activity, cry and consolability) score Behaviour 0 1 2 Face No particular expression or smile Occasional grimace or frown, withdrawn, disinterested Frequent to constant quivering chin, clenched jow Legs Normal position or relaxed Uneasy, restless, tense Kicking or legs drawn up Activity Lying quietly, normal position, moves easily Squirming, shifting, back and forth, tense Arched, rigid or jerking Cry No cry (awake or asleep) Moans or whimpers; occasional complaint Crying steadily, screams, sobs, frequent complaints Consolability Content, relaxed Reassured by touching, hugging or being talked to, distractible Difficult to console or comfort 0 = Relaxed and comfortable 1-3 = Mild discomfort 4-6 = Moderate pain 7-10 = Severe discomfort/pain
Postoperative revised FLACC scores | 8 hours postoperative
  Revised FLACC score ( face,leg,activity, cry and consolability) score Behaviour 0 1 2 Face No particular expression or smile Occasional grimace or frown, withdrawn, disinterested Frequent to constant quivering chin, clenched jow Legs Normal position or relaxed Uneasy, restless, tense Kicking or legs drawn up Activity Lying quietly, normal position, moves easily Squirming, shifting, back and forth, tense Arched, rigid or jerking Cry No cry (awake or asleep) Moans or whimpers; occasional complaint Crying steadily, screams, sobs, frequent complaints Consolability Content, relaxed Reassured by touching, hugging or being talked to, distractible Difficult to console or comfort 0 = Relaxed and comfortable 1-3 = Mild discomfort 4-6 = Moderate pain 7-10 = Severe discomfort/pain
Postoperative revised FLACC scores | 10 hours postoperative
  Revised FLACC score ( face,leg,activity, cry and consolability) score Behaviour 0 1 2 Face No particular expression or smile Occasional grimace or frown, withdrawn, disinterested Frequent to constant quivering chin, clenched jow Legs Normal position or relaxed Uneasy, restless, tense Kicking or legs drawn up Activity Lying quietly, normal position, moves easily Squirming, shifting, back and forth, tense Arched, rigid or jerking Cry No cry (awake or asleep) Moans or whimpers; occasional complaint Crying steadily, screams, sobs, frequent complaints Consolability Content, relaxed Reassured by touching, hugging or being talked to, distractible Difficult to console or comfort 0 = Relaxed and comfortable 1-3 = Mild discomfort 4-6 = Moderate pain 7-10 = Severe discomfort/pain
Postoperative revised FLACC scores | 12 hours postoperative
  Revised FLACC score ( face,leg,activity, cry and consolability) score Behaviour 0 1 2 Face No particular expression or smile Occasional grimace or frown, withdrawn, disinterested Frequent to constant quivering chin, clenched jow Legs Normal position or relaxed Uneasy, restless, tense Kicking or legs drawn up Activity Lying quietly, normal position, moves easily Squirming, shifting, back and forth, tense Arched, rigid or jerking Cry No cry (awake or asleep) Moans or whimpers; occasional complaint Crying steadily, screams, sobs, frequent complaints Consolability Content, relaxed Reassured by touching, hugging or being talked to, distractible Difficult to console or comfort 0 = Relaxed and comfortable 1-3 = Mild discomfort 4-6 = Moderate pain 7-10 = Severe discomfort/pain
Postoperative revised FLACC scores | 15 hours postoperative
  Revised FLACC score ( face,leg,activity, cry and consolability) score Behaviour 0 1 2 Face No particular expression or smile Occasional grimace or frown, withdrawn, disinterested Frequent to constant quivering chin, clenched jow Legs Normal position or relaxed Uneasy, restless, tense Kicking or legs drawn up Activity Lying quietly, normal position, moves easily Squirming, shifting, back and forth, tense Arched, rigid or jerking Cry No cry (awake or asleep) Moans or whimpers; occasional complaint Crying steadily, screams, sobs, frequent complaints Consolability Content, relaxed Reassured by touching, hugging or being talked to, distractible Difficult to console or comfort 0 = Relaxed and comfortable 1-3 = Mild discomfort 4-6 = Moderate pain 7-10 = Severe discomfort/pain
Postoperative revised FLACC scores | 18 hours postoperative
  Revised FLACC score ( face,leg,activity, cry and consolability) score Behaviour 0 1 2 Face No particular expression or smile Occasional grimace or frown, withdrawn, disinterested Frequent to constant quivering chin, clenched jow Legs Normal position or relaxed Uneasy, restless, tense Kicking or legs drawn up Activity Lying quietly, normal position, moves easily Squirming, shifting, back and forth, tense Arched, rigid or jerking Cry No cry (awake or asleep) Moans or whimpers; occasional complaint Crying steadily, screams, sobs, frequent complaints Consolability Content, relaxed Reassured by touching, hugging or being talked to, distractible Difficult to console or comfort 0 = Relaxed and comfortable 1-3 = Mild discomfort 4-6 = Moderate pain 7-10 = Severe discomfort/pain
Postoperative revised FLACC scores | 21 hours postoperative
  Revised FLACC score ( face,leg,activity, cry and consolability) score Behaviour 0 1 2 Face No particular expression or smile Occasional grimace or frown, withdrawn, disinterested Frequent to constant quivering chin, clenched jow Legs Normal position or relaxed Uneasy, restless, tense Kicking or legs drawn up Activity Lying quietly, normal position, moves easily Squirming, shifting, back and forth, tense Arched, rigid or jerking Cry No cry (awake or asleep) Moans or whimpers; occasional complaint Crying steadily, screams, sobs, frequent complaints Consolability Content, relaxed Reassured by touching, hugging or being talked to, distractible Difficult to console or comfort 0 = Relaxed and comfortable 1-3 = Mild discomfort 4-6 = Moderate pain 7-10 = Severe discomfort/pain
Postoperative revised FLACC scores | 24 hours postoperative
  Revised FLACC score ( face,leg,activity, cry and consolability) score Behaviour 0 1 2 Face No particular expression or smile Occasional grimace or frown, withdrawn, disinterested Frequent to constant quivering chin, clenched jow Legs Normal position or relaxed Uneasy, restless, tense Kicking or legs drawn up Activity Lying quietly, normal position, moves easily Squirming, shifting, back and forth, tense Arched, rigid or jerking Cry No cry (awake or asleep) Moans or whimpers; occasional complaint Crying steadily, screams, sobs, frequent complaints Consolability Content, relaxed Reassured by touching, hugging or being talked to, distractible Difficult to console or comfort 0 = Relaxed and comfortable 1-3 = Mild discomfort 4-6 = Moderate pain 7-10 = Severe discomfort/pain
Total postoperative paracetamol | one day after surgery
total postoperative Ketorolac | one day after surgery
number of participants developed complications | one day after operation
The satisfaction of the parents about the postoperative analgesia | 24 hours after surgery
  parent satisfaction score 1= very unsatisfied 2=unsatisfied 3= satisfied 4= very satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Abassia, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes